CLINICAL TRIAL: NCT06375148
Title: A Questionnaire Survey on Cognition of Enteral Nutrition Implementation in Patients Requiring Mechanical Ventilation in Prone Position
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Yan2024-0052
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Enteral Nutrition; Prone Position
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Zhejiang Quality Control Center
  Interventions: Other: Enteral nutrition
- Sichuan Provincial Center for quality control of TCM critical care medicine
  Interventions: Other: Enteral nutrition
- Severe nutrition group / nursing group of Zhejiang nutrition branch
  Interventions: Other: Enteral nutrition
- Critical care medicine of China Research Hospital Association
  Interventions: Other: Enteral nutrition

INTERVENTIONS:
Other: Enteral nutrition — prone position ventilation

SUMMARY:
Prone ventilation is an important treatment for respiratory failure with intractable hypoxia, and the Corona Virus Disease 2019(COVID-19 ) outbreak has further elevated the status of prone ventilation. Early enteral nutrition (EN) is also recognised as an important measure to improve the prognosis of critically ill patients. However, the administration of enteral nutrition during prone position is still quite controversial. In this paper, we analysed the tolerance and safety of enteral nutrition in the prone position by reviewing studies before and after the COVID-19 outbreak. Key strategies to improve the tolerability of enteral nutrition in the prone position are also summarised and discussed.

DETAILED DESCRIPTION:
We plan to carry out the following research: through multi center investigation and research, to understand the current situation of critical care workers' cognition of enteral nutrition in patients with severe prone position ventilation. 1. research purpose: to understand the current situation of cognition of critically ill medical staff on enteral nutrition in patients with severe prone position ventilation. 2. research design and methods: This study includes three parts: 1. confirmation of the research object; 2. research content and specific content of the questionnaire; 3. statistical analysis of questionnaire results. Research object: investigation unit: intensive care unit (ICU) of secondary grade A and above comprehensive hospitals (including traditional Chinese medicine and integrated traditional Chinese and Western medicine hospitals), including comprehensive ICU, central ICU, emergency ICU, medical ICU, surgical ICU, brain ICU, and other specialized ICUs. respondents: medical staff working in the above ICU during the survey. It does not include resident trainees, interns and other types of personnel who are not in the Department. Refresher trainees, if their job is ICU medical care, can also fill in the questionnaire, but it should be noted that the unit filling in is the original unit, not the refresher unit. Research content: Investigation on the current situation of medical staff's understanding of enteral nutrition in patients with severe prone position ventilation: a multicenter investigation. The questionnaire is divided into three parts (basic information, prone position ventilation information, enteral nutrition). See the questionnaire for details. The main purpose is to describe the current situation of critical care physicians' cognition of the implementation of enteral nutrition in prone position requiring mechanical ventilation. The main outcome measure was whether enteral nutrition had been started before prone position, and whether enteral nutrition would be cut off because of the need for prone position. Research methods: for the research objects that meet the inclusion criteria, the electronic questionnaire was issued in January 2023 for questionnaire survey, and the electronic questionnaire data were exported in the background in February 2023, and the questionnaire data were sorted out for statistical analysis. The main ways to issue questionnaires are as follows: 1. issue questionnaires through the quality control center of Zhejiang Province; 2. the questionnaire was distributed through the quality control center of traditional Chinese medicine critical care medicine in Sichuan Province; 3. through the severe nutrition group / nursing group of Zhejiang nutrition branch; 4. the questionnaire was distributed through the critical care medicine branch of the Chinese Research Hospital Association; 5. through the emergency world and emcrit wechat platform; 6. other ways.

ELIGIBILITY:
Inclusion Criteria:

* The intensive care unit (ICU) of the secondary grade A and above general hospitals (including traditional Chinese medicine and integrated traditional Chinese and Western medicine hospitals), including comprehensive ICU, central ICU, emergency ICU, internal medicine ICU, surgical ICU, brain ICU, and other specialized ICUs.

Exclusion Criteria:

* Resident trainees, interns and other types of personnel not in the Department

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical staff working in the above ICU during the survey.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
A questionnaire survey on cognition of enteral nutrition implementation in patients requiring mechanical ventilation in prone position | The questionnaire method was started in April, and the data statistics were completed in June
  Questionnaires were sent out in April, and data statistics were carried out in June

CONTACTS AND LOCATIONS:
Overall Officials: Libing Jiang, MASTER, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University; Chengfei Wang, MASTER, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Shanxiang Xu, MASTER, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Yongan Xu, DOCTOR, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Zhenjiang, China

IPD SHARING:
Plan to Share IPD: No